CLINICAL TRIAL: NCT04603976
Title: Registry for Migraine - Clinical Core
Acronym: REFORM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Messoud Ashina, Professor of Neurology, Danish Headache Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20019411
Record Dates: First submitted 2020-10-07; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — erenumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Arm (Experimental): Erenumab packed in a SureClick® Autoinjector Pen (AI)
  Interventions: Drug: Erenumab

INTERVENTIONS:
Drug: Erenumab — Erenumab 70 mg or 140 mg packed in a SureClick® Autoinjector Pen (AI)
  Other Names: Aimovig

SUMMARY:
This study aims to investigate the effect of erenumab on efficacy outcomes, tolerability outcomes, and patient-reported outcomes in individuals with migraine. Furthermore, the study aims to identify clinical predictors of erenumab response.

DETAILED DESCRIPTION:
Migraine is a prevalent neurological disorder and a leading cause of years lived with disability worldwide. As of recent, therapies targeting calcitonin gene-related peptide (e.g. erenumab) have been approved for the preventive treatment of migraine. This study aims to investigate the effect of erenumab on efficacy outcomes, tolerability outcomes, and patient-reported outcomes in individuals with migraine. Furthermore, the study aims to identify clinical predictors of erenumab response.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study-specific activities/procedures
* Age greater than or equal to 18 years upon entry into screening
* History of migraine (with or without aura) for greater than or equal to 12 months before screening according to the International Headache Society (IHS) Classification ICHD-3 (Headache Classification Committee of the International Headache Society, 2018) based on medical records and/or patient self report
* Greater than or equal to 4 headache days that meet criteria as migraine days per month on average across the 3 months before screening after baseline period
* Must have demonstrated greater than or equal to 75% compliance in headache diiary usage during baseline period

Exclusion Criteria:

Subjects are excluded from the study if any of the following criteria apply:

Disease Related

* Greater than 50 years of age at migraine onset
* History of cluster headache or hemiplegic migraine headache
* Inability to differentiate between migraine from other headaches
* The subject is at risk of self-harm or harm to others as evidenced by past suicidal behaviour
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator would pose a risk to subject safety or interfere with the study evaluation, procedures or completion Prior/Concomitant Therapy
* Previously received erenumab (Aimovig®)
* Received an anti-CGRP monoclonal antibody within 3 months prior to the start of the baseline period Prior/Concurrent Clinical Study Experience
* Currently receiving treatment in another investigational device or drug study, or less than 30 days or 5 half-lives since ending treatment on another investigational device or drug study (ies). Other investigational procedures while participating in this study are excluded.

Other Exclusions

* Female subjects of childbearing potential with a positive pregnancy test assessed at screening or day 1 by a urine pregnancy test.
* Female subject is pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 16 weeks after the last dose of investigational product.
* Female subjects of childbearing potential unwilling to use 1 acceptable method of effective contraception during treatment and for an additional 16 weeks after the last dose of investigational product.
* Evidence of current pregnancy or breastfeeding per subject self-report or medical records
* Subject has known sensitivity to any of the products or components to be administered during dosing
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the subject and investigator's knowledge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-09-25 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Headache Diary | Baseline Phase (Day -28 to Day 1) to Week 24
  Headache diary with daily entries to record migraine-related data.

SECONDARY OUTCOMES:
Headache Diary | Baseline Phase (Day -28 to Day 1) to Week 48
  Headache diary with daily entries to record migraine-related data.
Semi-Structured Interview | Screening Visit (Day -28)
  In-person semi-structured interview to record migraine-related data.
Headache Impact Test (HIT-6) | Baseline Phase (Day -28 to Day 1) to Week 24
  6-item questionnaire to assess headache-related disability
Headache Impact Test (HIT-6) | Baseline Phase (Day -28 to Day 1) to Week 48
  6-item questionnaire to assess headache-related disability
Migraine Disability Assessment Test (MIDAS) | Baseline Phase (Day -28 to Day 1) to Week 24
  7-item questionnaire to assess migraine-related disability
Migraine Disability Assessment Test (MIDAS) | Baseline Phase (Day -28 to Day 1) to Week 48
  7-item questionnaire to assess migraine-related disability
Hospital Anxiety and Depression Scale (HADS) | Baseline Phase (Day -28 to Day 1) to Week 24
  14-item questionnaire to assess anxiety and depression
Hospital Anxiety and Depression Scale (HADS) | Baseline Phase (Day -28 to Day 1) to Week 48
  14-item questionnaire to assess anxiety and depression
Pittsburgh Sleep Quality Index (PSQI) | Baseline Phase (Day -28 to Day 1) to Week 24
  19-item questionnaire to assess quality of sleep
Pittsburgh Sleep Quality Index (PSQI) | Baseline Phase (Day -28 to Day 1) to Week 48
  19-item questionnaire to assess quality of sleep
12-item Allodynia Symptom Checklist (ASC-12) | Baseline Phase (Day -28 to Day 1) to Week 24
  12-item questionnaire to allodynia
12-item Allodynia Symptom Checklist (ASC-12) | Baseline Phase (Day -28 to Day 1) to Week 48
  12-item questionnaire to allodynia
WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) | Baseline Phase (Day -28 to Day 1) to Week 24
  Questionnaire to assess health status and disability
WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) | Baseline Phase (Day -28 to Day 1) to Week 48
  Questionnaire to assess health status and disability
Neck Disability Index (NDI) | Baseline Phase (Day -28 to Day 1) to Week 24
  Questionnaire to assess neck disability
Neck Disability Index (NDI) | Baseline Phase (Day -28 to Day 1) to Week 48
  Questionnaire to assess neck disability
Low Back Pain Disability Questionnaire | Baseline Phase (Day -28 to Day 1) to Week 24
  Questionnaire to assess low back pain disability
Low Back Pain Disability Questionnaire | Baseline Phase (Day -28 to Day 1) to Week 48
  Questionnaire to assess low back pain disability

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, MD, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark

REFERENCES:
- [Derived] Thuraiaiyah J, Christensen RH, Al-Khazali HM, Wiggers A, Ashina M, Ashina H. Overlap between perceived triggers, premonitory symptoms and symptom persistence across migraine phases: A REFORM study. Cephalalgia. 2025 Aug;45(8):3331024251364234. doi: 10.1177/03331024251364234. Epub 2025 Aug 26. PMID 40980937
- [Derived] Karlsson WK, Christensen RH, Al-Khazali HM, Kallemose T, Jawad BN, Andersen O, Ashina M, Ashina H. Plasma SuPAR and therapeutic response to erenumab in migraine: a REFORM study. J Headache Pain. 2025 Apr 24;26(1):86. doi: 10.1186/s10194-025-02037-9. PMID 40275185
- [Derived] Karlsson WK, Ashina H, Cullum CK, Christensen RH, Al-Khazali HM, Amin FM, Ashina M; REFORM Investigators. The Registry for Migraine (REFORM) study: methodology, demographics, and baseline clinical characteristics. J Headache Pain. 2023 Jun 12;24(1):70. doi: 10.1186/s10194-023-01604-2. PMID 37303034